CLINICAL TRIAL: NCT01316302
Title: A 12-Week Double-Blind, Placebo-Controlled, Flexible-Dose Trial of Pristiq® (Desvenlafaxine) Extended-Release Tablets in Generalized Social Anxiety Disorder
Brief Title: 12-Week Study of Pristiq (Desvenlafaxine) Social Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Medical Research Network (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PF2010SAD; WS1228302 (Other Grant/Funding Number: Pfizer, Inc.)
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Social Phobia; SAD
MeSH Terms: conditions — Phobia, Social | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pristiq (Experimental): Flexible dose, 50-100mg QD
  Interventions: Drug: Pristiq
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pristiq — Flexible dose, 50-100mg QD, for 12 weeks.
  Other Names: desvenlafaxine
  Arms: Pristiq
Drug: Placebo — Matching placebo, taken QD for 12 weeks.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of Pristiq® in treatment of the symptoms of Generalized Social Anxiety Disorder (SAD).

DETAILED DESCRIPTION:
Social Anxiety Disorder (SAD) is recognized as a prevalent, chronic and disabling condition. Lifetime prevalence has been estimated at 13% in the National Comorbidity Survey. There is good reason to think that Pristiq® would be effective in Social Anxiety Disorder. Effexor XR, which is mechanistically similar to Pristiq®, was found effective for subjects with Generalized Social Anxiety Disorder in all five of the placebo controlled trials in which it was studied.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give written informed consent prior to any study procedures.
* Diagnosis of Social Anxiety Disorder (SAD) (300.23 Social Phobia/Social Anxiety Disorder, Generalized Subtype) according to DSM-IV-TR criteria, as determined by psychiatric evaluation with the Principal Investigator.
* A minimum score of 60 on the LSAS total score at both Screening and Baseline visits.
* A total HAM-D score of less than 15 at the Screening visit.
* CGI Severity score of 4 or greater at both Screening and Baseline visits.
* Female subjects of childbearing potential must commit to an effective form of contraception for the duration of the trial. Effective forms of contraception include: condoms with spermicide, diaphragm with spermicide, hormonal contraceptive agents (oral, transdermal, or injectable), and implantable contraceptive devices.

Exclusion Criteria:

* An Axis I disorder other than SAD (e.g., post-traumatic stress disorder, obsessive compulsive disorder, panic disorder) within 24 weeks of the Baseline visit. Subjects with co-morbid MDD, GAD, dysthymia, or specific phobias will be allowed if GSAD is the primary disorder in terms of clinical severity, as determined by the investigator.
* Any history or complication of schizophrenia or bipolar disorder.
* Any complication of body dysmorphic disorder.
* Substance dependence, as defined by DSM-IV-TR criteria, within 24 weeks of the Baseline visit.
* Subjects who are currently pregnant, lactating, or of childbearing potential and not practicing an effective method of contraception.
* Subjects scoring >2 on item #3 of the HAM-D, or who, in the opinion of the PI, are at a clinically significant risk for suicide.
* Systolic blood pressure ≥165 and/or diastolic blood pressure ≥95.
* Positive Urine Drug Screen at the Screening visit.
* Any current unstable and/or clinically significant medical condition, based on history or as evidenced in Screening laboratory and ECG assessments.
* Any history or complication of cancer or malignant tumor.
* Fluoxetine within 28 days of Baseline
* MAO inhibitors within 14 days of Baseline - Any other psychotropics (including SSRIs, SNRIs, and benzodiazepines) within 14 days of Baseline. Zolpidem (Ambien®) PRN is allowed for insomnia if not taken more than 3 times per week.
* Subjects who started psychotherapy or cognitive-behavioral therapy within 24 weeks of the Baseline visit, except for supportive psychotherapy.
* Electro-convulsive therapy (ECT) within 12 weeks of the Baseline visit.
* Treatment refractory GSAD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Liebowitz, MD, Principal Investigator — The Medical Research Network
Locations (1):
- The Medical Research Network, LLC, New York, New York, United States

REFERENCES:
- See also: Click here for more information about The Medical Research Network. — http://www.MedicalResearchNetwork.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pristiq | Placebo
Started | 30 | 33
Completed | 20 | 22
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pristiq | Placebo | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (14.6) | 41.9 (13.7) | 40.0 (19.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 33 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 14 | 20 | 34
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in the Liebowitz Social Anxiety Scale (LSAS) Total Score
Description: Liebowitz Social Anxiety Scale, measuring social anxiety symptoms; possible total scores ranging from 0-144, with higher scores indicating greater severity of symptoms.
Time Frame: Baseline to study endpoint (Week 12)
Population: The number of participants for analysis was 29 subjects per arm; data analyzed at Week 12 or Last Observation Carried Forward for the 16 subjects who dropped out before completion. Five other randomized subjects (1 on drug, 4 on placebo) were excluded from the ITT sample because of insufficient data (n = 4) or poor compliance (n = 1).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pristiq | Placebo
Number analyzed (Participants) | 29 | 29
Scores on a scale
  Mean baseline LSAS total | 93.4 (17.1) | 92.1 (16.8)
  Endpoint LSAS total | 55.0 (27.4) | 63.4 (22.1)
  Mean LSAS change from baseline | 38.4 (28.8) | 28.7 (24.2)

2. Secondary Outcome: Clinical Global Impression of Improvement Scale (CGI-I)
Description: CGI-I: one item, measuring overall improvement of illness; possible scores range from 1-7, with lower scores representing greater improvement. CGI-I responders: defined as having a CGI-I scores of 1 or 2 at Week 12/study endpoint.
Time Frame: Baseline to Week 12
Measure: Number; unit: % of subjects who were CGI-I responders
Arm/Group | Pristiq | Placebo
Number analyzed (Participants) | 29 | 29
% of subjects who were CGI-I responders | 69 | 48.3

3. Secondary Outcome: Patient Global Impression of Change
Description: Subject-rated global outcome scale. Subjects who rated themselves as 1 (Very Much Improved) or 2 (Much Improved) on the PGIC were considered self-rated responders.
Time Frame: Baseline to study endpoint (Week 12)
Measure: Number; unit: percentage of self-rated responders
Arm/Group | Pristiq | Placebo
Number analyzed (Participants) | 29 | 29
percentage of self-rated responders | 44.8 | 40.7

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Pristiq | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 26/30 | 25/33
OTHER ADVERSE EVENTS (reported when occurring in more than .06% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pristiq (N=30) | Placebo (N=33)
dizziness/lightheadedness/feeling faint (General disorders) | 11 (12) | 4 (6)
nausea/queasiness (General disorders) | 11 (16) | 3 (3)
drowsiness (General disorders) | 7 (9) | 2 (2)
insomnia (Nervous system disorders) | 5 (8) | 4 (4)
headache (General disorders) | 4 (6) | 5 (6)
fatigue (General disorders) | 4 (4) | 4 (5)
decreased appetite (General disorders) | 6 (7) | 1 (1)
indigestion (Gastrointestinal disorders) | 4 (4) | 1 (2)
flu/flu symptoms (General disorders) | 2 (2) | 3 (3)
soft stools/diarrhea (General disorders) | 5 (5) | 0 (0)
dry mouth (General disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No